CLINICAL TRIAL: NCT06472622
Title: Functional Neuroimaging to Detect the Neural Signatures of the Unpleasantness of Pain and Effort
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10001925; 001925-N
Record Dates: First submitted 2024-06-22; First posted 2024-06-25 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11-25

CONDITIONS: Fatigue Syndrome, Chronic
Keywords: Punishment; Fatigue Syndrome, Chronic; Pain; Physical Exertion; Effort; Brain; Magnetic Resonance Imaging; Neuroimaging; Psychophysics; Reward
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): This is a single-arm study. The order of intervention administration will be counterbalanced within this single arm.
  Interventions: Device: Thermal Pain Stimulation; Device: Physical Effort Stimulation

INTERVENTIONS:
Device: Thermal Pain Stimulation — Thermal pain will be administered during fMRI neuroimaging via a thermal stimulation device (Medoc Ltd., Advanced Medical System, Israel; 510K: K052357; K041908; K922052) to examine brain activity corresponding to the experience of this stimulus. This device and associated system carries an FDA 510 (K) clearance.
Device: Physical Effort Stimulation — Physical effort will be administered during fMRI neuroimaging via a hand dynamometer attachment for a physiological monitoring system (BIOPAC Systems, Inc., Goleta, CA, USA) to examine brain activity corresponding to the experience of this stimulus. This device has not received pre-marked approval or 510 (K) clearance by the FDA.

SUMMARY:
Background:

The way the brain processes rewards and punishments may play a role in some disorders of the nervous system. People with chronic overlapping pain conditions (such as myalgic encephalomyelitis/chronic fatigue syndrome [ME/CFS]) may have heightened responses to unpleasant, punishing sensations. Some of these conditions may also cause heightened responses to effort; this is an unpleasant sensation felt during physical and mental exertion.

Objective:

To learn more about how the brain processes different unpleasant sensations.

Eligibility:

People aged 18 to 50 years with ME/CFS. Healthy volunteers are also needed.

Design:

Participants will have 3 visits in 1 to 5 weeks.

Visit 1: Participants may have a neurologic exam. They will have a mock magnetic resonance imaging (MRI) scan. They will lie on a bed in a wooden tube while they practice 2 tasks:

Thermal pain rating: A device that creates mild to moderate heat will be placed on one leg.

Physical effort rating: Participants will squeeze a plastic bar with different levels of force.

Visit 2: Participants will have a real MRI scan. They will lie on a table that slides into a large tube.

Visit 3: Participants will have another MRI scan. They will repeat the thermal pain and physical effort tasks while in the scanner. Sensors will be placed on 1 arm to measure how the muscles function as they squeeze the bar.

Their heart rate will be tested: They will hold their finger against a camera lens for 1 minute. They will do 2 other tasks: 1 requires repeatedly pressing a key on a keyboard, and the other requires squeezing a bar.

DETAILED DESCRIPTION:
Study Description:

This protocol will examine the associations between brain activation and the subjective unpleasantness associated with pain and physical effort in healthy individuals. We have developed two behavioral tasks for administration during neuroimaging: a Thermal Pain Rating task and a Physical Effort Rating task, which will allow us to identify brain regions in which activity is associated with the unpleasantness of these experiences. We hypothesize that the unpleasantness of the experiences will be associated with activity in a recently identified network of brain regions thought to be involved in computing subjective value, known as the subjective valuation network (SVN).

Objectives:

Primary Objectives:

1. Determine which regions of the SVN are specifically involved in the subjective experience of unpleasantness associated with sensations of pain.
2. Determine which regions of the SVN are specifically involved in the subjective experience of unpleasantness associated with sensations of physical effort.

Endpoints:

Primary Endpoints:

1. SVN regions in which activity is significantly associated with unpleasantness of pain.
2. SVN regions in which activity is significantly associated with unpleasantness of physical effort.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy Controls: In order to be eligible to participate in this study as a healthy control, an individual must meet all the following criteria:

1. Ability of subject to understand and the willingness to sign a written informed consent document.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged 18-50 (inclusive).
4. Good general health as evidenced by medical history and/or physical examination.

ME/CFS Patients: In order to be eligible to participate in this study as an ME/CFS patient, an individual must meet all the following criteria:

1. Ability of subject to understand and the willingness to sign a written informed consent document.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged 18-50 (inclusive).
4. Has a diagnosis of ME/CFS, meeting at least one of three ME/CFS criteria: the 1994 Fukuda Criteria, the 2003 Canadian Consensus Criteria for Myalgic Encephalomyelitis/Chronic Fatigue Syndrome, or the Institute of Medicine Diagnostic Criteria.

EXCLUSION CRITERIA:

Healthy Controls:

1. Any current major neurological or psychiatric disorder such as (but not limited to) stroke, Parkinson s disease, Alzheimer s disease, schizophrenia, or major depressive disorder.
2. Any other current major medical disorder, such as a kidney disease, liver disease, cardiovascular disease, chronic pain condition, or any other disorder which, in the opinion of the PI would make participation risky for the individual or negatively affect the individual s ability to cooperate with study procedures.
3. Current use of medications acting primarily on the central nervous system, such as antidepressants, stimulants, etc.
4. Use of opioid medications for more than two weeks within the last two years or any use in the last month.
5. Current or history of substance use disorder, binge drinking, illegal drug use, or excessive tobacco use (defined as more than 10 cigarettes of nicotine per week).
6. Any more than occasional use of cannabis, defined as a score >1 (indicating use on more than one or two days in the last two weeks) on the marijuana use item of the DSM-5 Level 2-Substance Use-Adult questionnaire.
7. Any use of other illicit drugs or misuse of prescription medications, defined as a score >0 on any of the other items of the DSM-5 Level 2-Substance Use-Adult questionnaire.
8. Condition or injury affecting grip.
9. Condition or injury affecting extremities that would alter peripheral sensitivity to painful thermal stimuli or would otherwise cause such stimuli to be contraindicated.
10. Contraindications to MRI, including ferromagnetic metal in the cranial cavity or eye, implanted neural stimulator, cochlear implant, or ocular foreign body, implanted cardiac pacemaker, auto-defibrillator, or pump, non-removable body piercing, claustrophobia, inability to lie supine for 90 minutes, known pregnancy, or plans to become pregnant during the study.
11. Members of the NINDS BNU and their family members.
12. Non-English speakers will be excluded from the study as several study instruments do not have validated translations.

ME/CFS Patients:

1. Any current major neurological or psychiatric disorder, other than ME/CFS, such as (but not limited to) stroke, Parkinson s disease, Alzheimer s disease, schizophrenia, or major depressive disorder.
2. Any other current major medical disorder, other than ME/CFS, such as a kidney disease, liver disease, cardiovascular disease, chronic pain condition, or any other disorder which, in the opinion of the PI would make participation risky for the individual or negatively

   affect the individual s ability to cooperate with study procedures.
3. Current use of psychomotor stimulants, antipsychotics, or benzodiazepines.
4. Use of opioid medications for more than two weeks within the last two years or any use in the last month.
5. Current or history of substance use disorder, binge drinking, illegal drug use, or excessive tobacco use (defined as more than 10 cigarettes of nicotine per week).
6. Any more than occasional use of cannabis, defined as a score >1 (indicating use on more than one or two days in the last two weeks) on the marijuana use item of the DSM-5 Level 2-Substance Use-Adult questionnaire.
7. Any use of other illicit drugs or misuse of prescription medications, defined as a score >0 on any of the other items of the DSM-5 Level 2-Substance Use-Adult questionnaire.
8. Condition or injury affecting grip.
9. Condition or injury affecting extremities that would alter peripheral sensitivity to painful thermal stimuli or would otherwise cause such stimuli to be contraindicated.
10. Contraindications to MRI, including ferromagnetic metal in the cranial cavity or eye, implanted neural stimulator, cochlear implant, or ocular foreign body, implanted cardiac pacemaker, auto-defibrillator, or pump, non-removable body piercing, claustrophobia, inability to lie supine for 90 minutes, known pregnancy, or plans to become pregnant during the study.
11. Members of the NINDS BNU and their family members.
12. Non-English speakers will be excluded from the study as several study instruments do not have validated translations.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2034-06-30 (Estimated); Study Completion 2034-06-30 (Estimated)

PRIMARY OUTCOMES:
Determine which regions of the SVN are specifically involved in the subjective experience of unpleasantness associated with sensations of pain. | The measurement will be assessed concurrently with thermal pain stimulus administration during the fMRI procedure associated with one of the study visits, 1-31 days following the visit for the first session.
  SVN regions in which activity is significantly associated with unpleasantness of pain.
Determine which regions of the SVN are specifically involved in the subjective experience of unpleasantness associated with sensations of physical effort. | The measurement will be assessed concurrently with physical effort stimulus administration during the fMRI associated with one of the study visits, 1-31 days following the visit for the first session.
  The SVN has been hypothesized to play a role in producing the unpleasantness of negative experiences including effort.

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Wassermann, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
It has not been determined if data analysis based on IPD is beneficial or feasible. This will be evaluated at a later time.

REFERENCES:
- [Background] Zald DH, Treadway MT. Reward Processing, Neuroeconomics, and Psychopathology. Annu Rev Clin Psychol. 2017 May 8;13:471-495. doi: 10.1146/annurev-clinpsy-032816-044957. Epub 2017 Mar 15. PMID 28301764
- [Background] Chong TT, Bonnelle V, Manohar S, Veromann KR, Muhammed K, Tofaris GK, Hu M, Husain M. Dopamine enhances willingness to exert effort for reward in Parkinson's disease. Cortex. 2015 Aug;69:40-6. doi: 10.1016/j.cortex.2015.04.003. Epub 2015 Apr 20. PMID 25967086
- [Background] Peters J, Buchel C. Overlapping and distinct neural systems code for subjective value during intertemporal and risky decision making. J Neurosci. 2009 Dec 16;29(50):15727-34. doi: 10.1523/JNEUROSCI.3489-09.2009. PMID 20016088
- [Background] Levy DJ, Glimcher PW. The root of all value: a neural common currency for choice. Curr Opin Neurobiol. 2012 Dec;22(6):1027-38. doi: 10.1016/j.conb.2012.06.001. Epub 2012 Jul 3. PMID 22766486
- [Background] Basten U, Biele G, Heekeren HR, Fiebach CJ. How the brain integrates costs and benefits during decision making. Proc Natl Acad Sci U S A. 2010 Dec 14;107(50):21767-72. doi: 10.1073/pnas.0908104107. Epub 2010 Nov 30. PMID 21118983
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001925-N.html